CLINICAL TRIAL: NCT00244933
Title: Phase II Trial of Gemcitabine and Genistein in Metastatic Breast Cancer Patients With Biomarker Assays
Brief Title: Gemcitabine Hydrochloride and Genistein in Treating Women With Stage IV Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Lawrence E. Flaherty, Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2597; P30CA022453 (NIH); WSU-C-2597 (Other: Barbara Ann Karmanos Cancer Institute)
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Results first posted 2015-02-02 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Genistein; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine, genistein (Novasoy), Tumor biopsy (Experimental): Gemcitabine IV-1000mg/m2: Days 1 & 8 every 21 days Novasoy Orally-100 mg 2 times/day for 7 days; 2 times/day on Days 1-21 every 21 days.
  Interventions: Dietary Supplement: genistein; Drug: gemcitabine; Procedure: Tumor biopsy

INTERVENTIONS:
Dietary Supplement: genistein — Novasoy Orally-100 mg 2 times/day for 7 days; 2 times/day on Days 1-21 every 21 days.
  Other Names: Novasoy
Drug: gemcitabine — Gemcitabine IV-1000mg/m2: Days 1 & 8 every 21 days
  Other Names: Gemcitabine hydrochloride; Gemzar®
Procedure: Tumor biopsy — Biopsy of tumor prior to dose of genistein (Novasoy)

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine hydrochloride and genistein, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving gemcitabine hydrochloride together with genistein may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving gemcitabine hydrochloride together with genistein works in treating women with stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the objective response rate in patients with stage IV breast cancer treated with gemcitabine hydrochloride and genistein.

Secondary

* Determine the duration of response and survival of patients treated with this regimen.
* Determine the time to disease progression in patients treated with this regimen.
* Determine the quantitative and qualitative toxic effects of this regimen in these patients.
* Correlate plasma genistein levels with response in patients treated with this regimen.

OUTLINE: Patients receive oral genistein once daily on days -7 to 1. Patients also receive gemcitabine hydrochloride IV on days 1 and 8 and oral genistein once daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 36 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed breast cancer

  * Stage IV disease
  * Clinical and/or radiological evidence of metastatic disease
* Measurable disease

  * Prior radiotherapy allowed provided there is ≥ 1 measurable disease site outside the radiation field
* No active CNS metastases

  * Previously treated CNS metastases allowed provided disease is stable for ≥ 3 months without steroids or antiseizure medications
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Sex

* Female

Menopausal status

* Not specified

Performance status

* SWOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10 g/dL

Hepatic

* Bilirubin ≤3.0 mg/dL
* AST and ALT ≤ 2.5 times upper limit of normal

Renal

* Creatinine ≤ 1.5 mg/dL

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No serious systemic disorder that would preclude study compliance
* No history of another malignancy except curatively treated carcinoma of the cervix or basal cell or squamous cell skin cancer in complete remission
* No unresolved bacterial infection requiring antibiotic treatment
* No known HIV-1 positivity

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 3 weeks since prior biologic therapy

Chemotherapy

* Prior adjuvant chemotherapy allowed
* Prior adjuvant or neoadjuvant taxane-based therapy or taxane therapy for metastatic disease allowed

  * Patient must have failed therapy within 2 years after completion of treatment
* At least 3 weeks since prior chemotherapy
* No more than 2 prior cytotoxic chemotherapy regimens for metastatic disease
* No prior gemcitabine hydrochloride
* No other concurrent chemotherapy

Endocrine therapy

* See Disease Characteristics
* At least 2 weeks since prior and no concurrent hormonal therapy

  * Must have documented disease progression during prior hormonal therapy

Radiotherapy

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy

Surgery

* At least 3 weeks since prior surgery

Other

* At least 3 weeks since prior investigational therapy
* At least 1 week since prior soy supplements (e.g., soy-based pills, liquids, or concentrates)

  * Dietary soy as part of a meal (e.g., tofu) allowed once a week
* No concurrent nutritional supplements, herbal agents, or high doses of antioxidants (e.g., vitamins C, D, or E) that may interact with, antagonize, alter, or imitate the potential effects of gemcitabine hydrochloride or genistein

  * A single daily multivitamin is allowed
* No other concurrent immunotherapy
* No other concurrent experimental medication
* Concurrent anticoagulants, appetite stimulants, and replacement steroids allowed

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2004-02; Primary Completion 2008-11 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Weise, DO, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gemcitabine, Genistein (Novasoy), Tumor Biopsy
Started | 19
Completed | 17
Not Completed | 2
Not completed — Not response evaluable | 2

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine, Genistein (Novasoy), Tumor Biopsy
Number analyzed (Participants) | 19
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 53 [31 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate by RECIST Criteria Following
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: every 2 courses until disease progression or death, up to 24 weeks
Measure: Number; unit: participants
Groups:
- Gemcitabine & Genistein: Gemcitabine, genistein (Novasoy), Tumor biopsy Gemcitabine IV-1000mg/m2: Days 1 & 8 every 21 days: Novasoy Orally-100 mg 2 times/day for 7 days; 2 times/day on Days 1-21 every 21 days.
Arm/Group | Gemcitabine & Genistein
Number analyzed (Participants) | 17
participants | 0

ADVERSE EVENTS:
Arm/Group | Gemcitabine & Genistein
Serious Adverse Events (participants affected / at risk) | 5/19
Other Adverse Events (participants affected / at risk) | 2/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine & Genistein (N=19)
White blood cells (WBC) (Investigations) | 5 (5)
Hemoglobin (Hgb) (Investigations) | 1 (1)
Absolute neutrophil count (ANC) (Investigations) | 5 (5)
Platelets (Investigations) | 3 (3)
Elevated Aspartate Aminotransferase (AST) (Investigations) | 1 (1)
Elevated Alanine Aminotransferase (ALT) (Investigations) | 1 (1)
Pain (General disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine & Genistein (N=19)
Hemoglobin (Hgb) (Investigations) | 1 (1)
Platelets (Investigations) | 1 (1)
Fatigue (General disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Elevated Alkaline Phosphate (Investigations) | 1 (1)
Pain (General disorders) | 2 (2)
Hot flashes (Vascular disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Although the study is designed to accrue 18 response evaluable participants in the first stage, the decision was made to close the study after 17 patients because of lack of efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2009-01-09): https://cdn.clinicaltrials.gov/large-docs/33/NCT00244933/Prot_SAP_000.pdf